CLINICAL TRIAL: NCT04709146
Title: The Influence of Covid-19 on the Audio-vestibular System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Yoni Evgeni Gutkovich, M.D/Ph.D., HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0226-20-EMC
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovered Covid-19 patients (Other): Diagnostic evulation with audiometry, Tympanography, SVV, VHIT, VNG.
  Interventions: Diagnostic Test: Audio-Vestibular evaluation
- Healthy Control (Other): Diagnostic evulation with audiometry, Tympanography, SVV, VHIT, VNG.
  Interventions: Diagnostic Test: Audio-Vestibular evaluation

INTERVENTIONS:
Diagnostic Test: Audio-Vestibular evaluation — Diagnostic evulation with audiometry, Tympanography, SVV, VHIT, VNG.

SUMMARY:
the study's porpuse is to examine whether Covid-19 causese a reduction in sensorineural hearing and vestibular function in recovered pateints - compared to healthy controls.

Both study groups will undergo audiometry, tympanometry, Video Head Impulse testing, Subjective Visual Vertigo testing and Video-Nystamography.

Previous audiometry results will also be aquired.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-80 performed audiometry testing in the last two years

Exclusion Criteria:

* known inner ear dysfunction - Sudden sensorineural hearing loss; autoimmune disease (Cogan's syndrom, SLE, ect.), familial/genetic sensorineural hearing loss, excessive noise exposure.

knowm conductive hearing loss (Air-bone gap>10dB) prior ear surgery chronic tympanic membrane perforation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
sensoneural hearing level - PTA | through study completion, an average of 1 year
  PTA at each frequency will be compared between new and baseline audiogram for each group. Afterwhich - the average PTA decreament would be compared betwenn both groups - contrl and recovered COVID-19 patients

SECONDARY OUTCOMES:
vestibular function | through study completion, an average of 1 year
  vestibular function will be compared netween the two groups after VHIT, SVV and VNG testing

IPD SHARING:
Plan to Share IPD: No